CLINICAL TRIAL: NCT04938635
Title: A Phase 2b, Double-blind, Randomised, Placebo-controlled, Multicentre Study to Assess the Efficacy and Safety of VIT-2763 Multiple Doses in Adults With Transfusion-dependent Beta-thalassaemia
Brief Title: Efficacy and Safety Study of Multiple Doses of VIT-2763 in Adults With Transfusion-dependent Beta-thalassemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic reasons
Sponsor: Vifor (International) Inc. (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIT-2763-THAL-203; 2021-001639-23 (EudraCT Number)
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-03

CONDITIONS: Beta-Thalassemia
Keywords: Beta-Thalassemia; Transfusion-dependent Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — VIT-2763; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VIT-2763 60 mg QD (Experimental): VIT-2763 60 mg administered once daily
  Interventions: Drug: VIT-2763 60 mg QD
- VIT-2763 60 mg BID (Experimental): VIT-2763 60 mg administered twice daily
  Interventions: Drug: VIT-2763 60 mg BID
- VIT-2763 120 mg BID (Experimental): VIT-2763 120 mg administered twice daily
  Interventions: Drug: VIT-2763 120 mg BID
- Placebo (Placebo Comparator): Placebo capsule administered twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIT-2763 60 mg QD — Participants receive one VIT-2763 60 mg capsule plus one Placebo capsule orally in the morning, and 2 Placebo capsules orally in the evening, for 24 weeks.
  Other Names: Vamifeport 60 mg QD
  Arms: VIT-2763 60 mg QD
Drug: VIT-2763 60 mg BID — Participants receive one VIT-2763 60 mg capsule plus one Placebo capsule orally, twice daily for 24 weeks.
  Other Names: Vamifeport 60 mg BID
  Arms: VIT-2763 60 mg BID
Drug: VIT-2763 120 mg BID — Participants receive two VIT-2763 60 mg capsules orally, twice daily for 24 weeks.
  Other Names: Vamifeport 120 mg BID
  Arms: VIT-2763 120 mg BID
Drug: Placebo — Participants receive two Placebo capsules matching VIT-2763 orally, twice daily for 24 weeks.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of 3 multiple doses of VIT-2763 as measured by the reduction in red blood cell (RBC) transfusion burden from Week 13 to Week 24, to identify the most efficacious and safe dose.

DETAILED DESCRIPTION:
All patients giving written informed consent will undergo a 12-week screening period to determine eligibility for study entry. At Day 1, patients who meet the eligibility requirements will be randomized in a double-blind manner to 1 of 4 treatment groups: VIT-2763 60 mg (once daily), 60 mg (twice daily), or 120 mg (twice daily) or placebo.

The randomisation will be stratified (balanced allocation across treatment groups) according to β0/β0 genotype (yes/no).

The duration of the treatment with VIT-2763 or placebo is 24 weeks, after which patients will undergo a 12-week post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥40.0 kg and ≤100 kg at screening
* Documented diagnosis of beta-thalassemia or Hb E/beta-thalassemia
* Red blood cell (RBC) transfusion dependence, defined as at least 6 RBC units in the 24 weeks prior to randomization and no transfusion-free period for ≥35 days during that period
* Ability to understand the requirements of the study and provide written informed consent

Exclusion Criteria:

* Documented diagnosis of Hb S/beta-thalassemia, alpha-thalassemia, or delta beta (δβ)-thalassemia, or hereditary persistence of foetal Hb.
* History of partial or total splenectomy within 4 months prior to screening.
* History of myocardial iron overload
* Chronic liver disease or history of liver cirrhosis
* Clinically relevant renal disease
* History or clinically important finding of cardiac disorders
* History of clinically significant lung disease
* Uncontrolled hypertension (> Grade 1 according to NCI CTCAE current version)
* Unable to take and absorb oral medications.
* Pregnancy or breastfeeding
* History of drug or alcohol abuse within 2 years prior to screening
* History or concomitant solid tumors and/or hematological malignancies unless resolved in the ≥5 past years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving ≥33% reduction of RBC transfusions from baseline and a reduction of ≥2 units assessed consecutively from Week 13 to Week 24 compared to the baseline transfusion | Week 13 to Week 24 comparing to Baseline (Day -83 to Day 1)

SECONDARY OUTCOMES:
Change from baseline in RBC transfusions over Weeks 13 to 24 compared to the baseline RBC transfusion burden derived using the last 12 weeks prior to randomization. | Week 13 to Week 24 comparing to Baseline (Day -83 to Day 1)
Proportion of patients achieving ≥50% reduction of RBC transfusions and ≥2 units assessed over any consecutive 12-week interval from Week 1 to 24. | Any consecutive 12-week interval from Week 1 to Week 24 comparing to Baseline (Day -83 to Day 1)
Proportion of patients achieving ≥33% reduction of RBC transfusions and ≥2 units assessed over any consecutive 12-week interval from Week 1 to 24. | Any consecutive 12-week interval from Week 1 to Week 24 comparing to Baseline (Day -83 to Day 1)
Mean change from baseline in Quality of Life (QoL) total score | Week 15 and Week 24 comparing to Baseline (Day 1)
  Transfusion-dependent QoL Questionnaire (TranQuol): a disease-specific, validated, QoL measure developed for thalassemia patients. The adult version includes 36 questions grouped into 5 domains: physical health, emotional health, sexual health, family functioning, and school/career functioning. The total score ranges from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szecsödy, Study Director — Vifor (International) Inc.
Locations (7):
- Investigator site #710, Whittier, California, United States
- Bulgaria (3):
  - Investigational site #802, Plovdiv
  - Investigational site #801, Sofia
  - Investigational site #804, Stara Zagora
- Israel (3):
  - Investigator Site 404, Jerusalem
  - Investigator Site 406, Petah Tikva
  - Investigator Site 405, Safed

IPD SHARING:
Plan to Share IPD: No